CLINICAL TRIAL: NCT04105439
Title: Relation Between Plasma Soluble Urokinase Plasminogen Activator Receptor and Behçet's Disease .
Brief Title: Plasma Soluble Urokinase Plasminogen Activator Receptor and Behçet's Disease .
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Farghaly Ramadan, resident doctor, Assiut University
Other Study IDs: suPAR in behcet disease
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Behçet Disease
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: healthy subjects who do not have the disease
- patients with Behçet's disease: subjects who do have the disease ( Behçet's disease )

SUMMARY:
The purpose of the study is to determine whether plasma levels of the soluble urokinase plasminogen activator(suPAR) can serve as a blood-based biomarker for diagnosis of Behçet's disease and its correlation with disease activity.

DETAILED DESCRIPTION:
Behçet's disease (BD) is a chronic, systemic vasculitis disease that can be evident in many systems and characterized by recurrent attacks, oral and/or genital aphthous ulcers, skin lesions, and inflammatory ocular findings. It was first described in 1937 by the Turkish dermatologist Hulusi Behçet.[1-3]

Although with an unclear pathogenesis, BD is considered a type of vasculitis triggered by immunological mechanisms. Increased levels of pro-inflammatory cytokines are reported in patients with BD. In the afflicted organs, a remarkable infiltration of neutrophils and lymphocytes can be seen.[4-6]

Diagnosis of BD is mainly clinical, on the association of symptoms, but diagnosis/classification criteria may help. Various sets of criteria were created for BD diagnosis and the recent one is the international criteria for Behçet's disease (ICBD) that was created by 27 countries in 2006 and revised in2014.[7]

There is no standard laboratory marker for the diagnosis and follow-up of BD. certain cytokines and increased serum levels of C-reactive protein (CRP) are considered as markers of disease activity.[8] Soluble urokinase plasminogen activator receptor (suPAR), a potential new biomarker, is a soluble form of the membrane-bound receptors expressed from and comprising mainly of various immune cells (monocytes, neutrophils, activated T lymphocytes, macrophages, endothelial cells, keratinocytes, smooth muscle cells and even tumor cells. [9] Numerous studies on various inflammatory diseases, cancer, tuberculosis, central nervous system infections, sepsis, liver fibrosis and inflammatory bowel disease have shown increased systemic levels of suPAR. In these diseases, suPAR systemic levels are shown to have a prognostic value in determining disease severity.[10]

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients diagnosed as Behçet's disease according to international study group criteria (ICBD ) for diagnosis of Behçet's

Exclusion Criteria:

* Age< 18 years
* Other autoimmune diseases.
* Pregnancy.
* Acute and chronic systemic infection history.
* The presence of chronic diseases such as chronic renal failure, liver and cardiac failure.
* Presence or history of cancer.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients age ≥ 18 years old and are diagnosed as Behçet's disease according to international study group criteria (ICBD ) for diagnosiss of Behçet's
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of the level of suPAR in the study subjects. | baseline
  to study the relation between leve of the marker and presence of the diesase.

SECONDARY OUTCOMES:
evaluation of the levels of suPAR with the activity of the disease. | baseline
  to study relation between level of the marker and activity of the disease

REFERENCES:
- [Background] Criteria for diagnosis of Behcet's disease. International Study Group for Behcet's Disease. Lancet. 1990 May 5;335(8697):1078-80. PMID 1970380
- [Background] Koc Y, Gullu I, Akpek G, Akpolat T, Kansu E, Kiraz S, Batman F, Kansu T, Balkanci F, Akkaya S, et al. Vascular involvement in Behcet's disease. J Rheumatol. 1992 Mar;19(3):402-10. PMID 1578454
- [Background] Kose O. Development of Immunopathogenesis Strategies to Treat Behcet's Disease. Patholog Res Int. 2012;2012:261989. doi: 10.1155/2012/261989. Epub 2012 Apr 3. PMID 22550612
- [Background] Tursen U. Pathophysiology of the Behcet's Disease. Patholog Res Int. 2012;2012:493015. doi: 10.1155/2012/493015. Epub 2011 Oct 1. PMID 21977335
- [Background] International Team for the Revision of the International Criteria for Behcet's Disease (ITR-ICBD). The International Criteria for Behcet's Disease (ICBD): a collaborative study of 27 countries on the sensitivity and specificity of the new criteria. J Eur Acad Dermatol Venereol. 2014 Mar;28(3):338-47. doi: 10.1111/jdv.12107. Epub 2013 Feb 26. PMID 23441863
- [Background] Adam B, Calikoglu E. Serum interleukin-6, procalcitonin and C-reactive protein levels in subjects with active Behcet's disease. J Eur Acad Dermatol Venereol. 2004 May;18(3):318-20. doi: 10.1111/j.1468-3083.2004.00907.x. PMID 15096143
- [Background] Gustafsson A, Ljunggren L, Bodelsson M, Berkestedt I. The Prognostic Value of suPAR Compared to Other Inflammatory Markers in Patients with Severe Sepsis. Biomark Insights. 2012;7:39-44. doi: 10.4137/BMI.S9460. Epub 2012 Apr 10. PMID 22550400
- [Background] Thuno M, Macho B, Eugen-Olsen J. suPAR: the molecular crystal ball. Dis Markers. 2009;27(3):157-72. doi: 10.3233/DMA-2009-0657. PMID 19893210
- See also: University of Leeds. Behçet's Disease Current Activity Form 2006. available at the site. — http://medhealth.leeds.ac.uk/download/910/behcetsdiseaseactivityform.